CLINICAL TRIAL: NCT00064454
Title: FACTS II: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-arm Study of the Efficacy and Safety of OPC-6535 Tablets in the Treatment of Subjects With Active Ulcerative Colitis
Brief Title: FACTS II: A Study to Test the Safety and Effectiveness of a New Medication on the Treatment of Active Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 197-02-218
Record Dates: First submitted 2003-07-08; First posted 2003-07-10 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — tetomilast; Pharmaceutical Preparations

INTERVENTIONS:
Drug: OPC-6535 Tablets (drug)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the drug OPC-6535 compared to a placebo in patients with active Ulcerative Colitis.

Depending on their response, participants will be offered the investigational medication for up to one year after the study's completion at select sites.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18-80 years of age, inclusive, who provide written informed consent prior to any study-related procedures and who are, in the opinion of the Investigator, likely to comply with all the requirements of the study
* Subjects with established diagnosis of active ulcerative colitis, who have relapsed within 12 weeks before screening. All subjects must have had the diagnosis of ulcerative colitis established by colonoscopy* prior to entering the study. (Newly diagnosed patients are also eligible.) * Colonoscopy may be substituted for flexible sigmoidoscopy during Screening if this inclusion criterion is not met.
* Colonic involvement with ulcerative colitis beyond 15 cm of the anal verge.
* Subjects with active disease, as defined by a DAI score between 7 and 11, inclusive, at the Screening/Baseline Visit.
* A score of ≥2 for rectal bleeding and a score ≥ 0 on flexible sigmoidoscopy at the Screening/Baseline Visit, based on DAI criteria.
* Subjects who have been on a stable dose of 5-ASA for at least 14 days prior to the Screening/Baseline Visit OR subjects who have not been receiving any 5-ASA for at least 14 days.
* Subjects who are surgically sterilized or who are prepared to and agree to practice a double-barrier form of birth control from the Screening/Baseline Visit through 30 (females) and 90 (males) days, respectively, from the last dose of study medication. Females who are more than 12 months post-menopausal are also eligible to participate in the study.

Exclusion Criteria:

* Subjects who have severe disease, defined as DAI of 12 at the Screening/Baseline Visit, and/or subjects whom the Investigator deems likely to require immunosuppressant therapy including corticosteroids and/or hospitalization during the period of study.
* Subjects who have any other clinically significant disease(s) which, in the opinion of the Investigator, could compromise the subject's involvement in the study and/or interfere with the absorption of the study drug or the overall interpretation of the data.
* Subjects who have had major gastrointestinal surgery including, but not limited to, a colostomy, an ileostomy or previous colonic surgery other than appendectomy.
* Subjects who have used oral corticosteroids (including oral budesonide) within 30 days, or topical intrarectal agents (corticosteroids or 5-ASA enemas, suppositories, foams) within 7 days of Screening/Baseline. (Topical dermatological corticosteroids are not excluded).
* Subjects who have used immunosuppressants including, but not limited to: azathioprine, 6-mercaptopurine, methotrexate, within 28 days or IL-10, IL-11, FK-506 [tacrolimus], mycophenolate, cyclosporine, anti-TNF-α or monoclonal antibody medications within 60 days of Screening/Baseline.
* Subjects who have a history of active malignancies within 5 years (surgically-treated basal cell, squamous cell, non-melanoma or in situ cervical carcinomas permissible), an intra-abdominal abscess, a toxic megacolon, or a clinical instability resulting from any other cause.
* Subjects with a known or suspected history of sclerosing cholangitis.
* Subjects with a known or suspected history of clinically relevant cardiac disease.
* Subjects with a positive stool culture for any enteric pathogens, pathogenic ova or parasites, or a positive EIA that is subsequently confirmed by a positive cytotoxin assay for C. difficile toxin. (Results for any enteric pathogens, pathogenic ova or parasites, but not C. difficile toxin, may be pending at the time of randomization and study drug initiation.)
* Subjects with a partial bowel obstruction, as documented by proximal small bowel dilation at Screening/Baseline.

Additional exclusion criteria apply. Please see study Web site for additional information.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375
Dates: Start 2003-05; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - Redpoint Research, Phoenix, Arizona
  - Desert Sun Gastroenterology, Tucson, Arizona
  - Central California Medical Research, Fresno, California
  - Rocky Mountain Clinical Research, Golden, Colorado
  - Gastroenterology Associated of Fairfield County, Bridgeport, Connecticut
  - Washington Fetterson, Washington Gastroenterology, Washington D.C., District of Columbia
  - Florida Medical Research Institute, Gainesville, Florida
  - Mark Lamet, Hollywood, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Bruce Salzberg, Atlanta, Georgia
  - Drug Research Services, Metairie, Louisiana
  - Metropolitan Gastroenterology Group, Chevy Chase, Maryland
  - Highland Medical Center, Braintree, Massachusetts
  - Minnesota Gastroenterology, Plymouth, Minnesota
  - Gastrointestial Associates, PA, Jackson, Mississippi
  - Affiliates in Gastroeneterology, Florham Park, New Jersey
  - Long Island Clinical Research Associates, LLP, Great Neck, New York
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - Charlotte Gastroenterology and Hepatology, Charlotte, North Carolina
  - Carolina Research Center, Greenville, North Carolina
  - Boice-Willis Clinic, Rocky Mount, North Carolina
  - West Hills Gastroenterology Associates, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Gastrointestinal Associates, Knoxville, Tennessee
  - Nashville Medical Research Institute, Nashville, Tennessee
  - System Endocrinology & Research Center, Houston, Texas
  - Internal Medicine Associates, Danville, Virginia
  - University of Wisconsin Medical School, Madison, Wisconsin